CLINICAL TRIAL: NCT04900389
Title: The Effect of Stigma, Anxiety and Wise Awareness Levels on Their Professional Lives With Respect to The Nurses' COVID-19 Status
Brief Title: The Effect of Nurses' Having COVID-19 on Their Professional Lives
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Gamze BULUT, Graduate student, Uludag University
Other Study IDs: 2021-4/49
Record Dates: First submitted 2021-05-14; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Stigma, Social; Anxiety
Keywords: Stigma; Anxiety; Wise awareness; COVID-19; Nurse
MeSH Terms: conditions — Social Stigma; Anxiety Disorders; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Nurses with COVID-19: The questionnaire form is included in the section on COVID-19. 2nd question; They will mark the answer "Yes" to the question "Have you been diagnosed with COVID-19?" 5th question; Individuals who answer "No" to the question "Have you been subjected to discriminatory behaviors by your environment because you were a healthcare worker during the COVID-19 pandemic process?" Will move on to the 11th question in the same section.
- Kontrol Group: Nurses who have not had COVID-19: The questionnaire form is included in the section on COVID-19. 2nd question; They will mark "No" to the question "Have you been diagnosed with COVID-19?" And move on to the 4th question in the same section.
  The 5th question in Annex 2 of the questionnaire form; Individuals who answer "No" to the question "Have you been subjected to discriminatory behaviors by your environment because you were a healthcare worker during the COVID-19 pandemic process?" Will move on to the 11th question in the same section.

SUMMARY:
Background: Since the first day of the epidemic, people diagnosed with COVID-19 and their relatives, some countries and groups such as healthcare professionals are exposed to discriminatory behavior and stigmatization in the world. Nurses fighting in the front lines from the very beginning of the epidemic and interacting with the patient the most experience anxiety and are exposed to stigma.

Aim: With this study, it was aimed to determine the stigma, anxiety and wise awareness levels of nurses in our country according to their COVID-19 experience and to determine their effect on their professional lives.

Methods: The universe of this case-control study, which will determine the level of stigma, anxiety and wise awareness of those who work as nurses in the clinic according to their COVID-19 passing status, is the universe of T.C. Nurses working at Ministry of Health Health Sciences University Bursa Yüksek İhtisas Training and Research Hospital Internal and Surgical Clinics (N: 756). The sample calculation of the research was calculated using the sampling method with known universe. The minimum number of people in the sample was calculated as (n) 354 when 1% error and 99% confidence interval were taken with the Raosoft sampling method. It was planned to reach the total number of nurses selected from internal and surgical clinics by using simple random sampling method and to collect data from these clinics between 15.05.2021 - 15.06.2021. In this study, socio-demographic information and questions about COVID-19, the Effect of COVID-19 Pandemic on Professional Life, "Coronavirus Anxiety Scale" and Toronto Wisdom Awareness Scale will be used in this study.

DETAILED DESCRIPTION:
Study Protocol, Methods and Procedures to be Applied The universe of this case-control study, which will determine the level of stigma, anxiety and wise awareness of those who work as nurses in the clinic according to their COVID-19 passing status, is the universe of T.C. Nurses working at Ministry of Health Health Sciences University Bursa Yüksek İhtisas Training and Research Hospital Internal and Surgical Clinics (N: 756). The sample calculation of the research was calculated using the sampling method with known universe. The minimum number of people in the sample was calculated as (n) 354 when 1% error and 99% confidence interval were taken with the Raosoft sampling method. It was planned to reach the total number of nurses selected from internal and surgical clinics by using simple random sampling method and to collect data from these clinics between 15.05.2021 - 15.06.2021. In this study, socio-demographic information and questions about COVID-19, the Effect of COVID-19 Pandemic on Professional Life, "Coronavirus Anxiety Scale" and Toronto Wisdom Awareness Scale will be used in this study. The part containing sociodemographic information is 11 questions. The section on COVID-19 is composed of 11 questions by literature review. The part of the effect of the COVID-19 Pandemic process on professional life is composed of 11 items (Participants will give points between 0 and 10 for the 1st, 2nd, 3rd and 9th items, 0: none, 10: quite often), (4th, 5th, Participants will score between 0 and 10 for the 6th, 7th, 8th, 10th and 11th items, 0: not at all, 10: quite a lot). Each item of the Coronavirus Anxiety Scale (CAS) is rated on a 5-point scale from 0 (not at all) to 4 (almost daily) based on experience over the past two weeks. A CAS total score of 9 indicates dysfunctional anxiety associated with coronavirus. High scores on a particular item or a high total scale score (9) may indicate problematic symptoms of the participant that may require further evaluation and / or treatment. Toronto Wisdom Awareness Scale (DPSS) consists of 13 items and a 5-Likert-type interval is used for each item (1: strongly disagree, 5: strongly agree). Scoring of the scale will be made according to the name of the factor. Scoring will be done in two separate groups as monitoring without being affected (Items 1, 2, 4, 7, 8, 9, 11) and Curiosity (Items 3, 5, 6, 10, 12, 13). Permission was obtained from the responsible authors who made the validity and reliability of the scales to be used in our study. The survey was conducted by researcher, T.C. The Ministry of Health Health Sciences University Bursa Yüksek İhtisas Training and Research Hospital will be held with nurses working in internal and surgical clinics. Due to the COVID-19 pandemic, the questionnaire form will be given to the nurses working in the clinic for application and will be taken back after a certain period of time. The Coronavirus Anxiety Scale and Toronto Wisdom Awareness Scale will also be included in the continuation of the questionnaire. Participants will score 5 items in CAS from 0 (not at all) to 4 (almost every day). Participants will give points to the items in the TBFÖ as 1: absolutely disagree, 2: disagree, 3: undecided, 4: agree, 5: absolutely agree. The total time is 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* T.R. Working as a Clinical (Internal and Surgical) Nurse at the Ministry of Health Health Sciences University Bursa High Specialization Training and Research Hospital,
* Agreeing to participate in the research voluntarily,
* Not having any visual, auditory and psychological problems that would hinder conducting surveys and scales,
* Be 18 years or older,
* At least high school graduate.

Exclusion Criteria:

* T.R. Not working as a Clinical (Internal and Surgical) Nurse at the Ministry of Health Health Sciences University Bursa High Specialization Training and Research Hospital,
* Refusing to voluntarily participate in the research,
* Having any visual, auditory and psychological problems that prevent making surveys and scales,
* Being under the age of 18,
* Not having at least a high school graduate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The universe of work T.C. Nurses working at Ministry of Health Health Sciences University Bursa Yüksek İhtisas Training and Research Hospital Internal and Surgical Clinics (N: 756). The sample calculation of the study was calculated using the sampling method with known universe. The minimum number of people required in the sample was calculated as (n) 354 when 1% error and 99% confidence interval were taken with the Raosoft sampling method. Reaching the total number of nurses selected from internal and surgical clinics by using simple random sampling method.
Sampling Method: Probability Sample
Enrollment: 354 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety levels of nurses according to their COVID-19 passing status | 5 months
  The Coronavirus Anxiety Scale (CAS) will be used. Each item of CAS is rated on a 5-point scale from 0 (not at all) to 4 (almost daily) based on experience over the past two weeks. A CAS total score of 9 indicates dysfunctional anxiety associated with coronavirus. High scores on a particular item or a high total scale score (9) may indicate problematic symptoms of the individual that may require further evaluation and / or treatment.

SECONDARY OUTCOMES:
Wise awareness levels of nurses based on their COVID-19 passing status | 5 months
  The Toronto Wisdom Awareness Scale (PACS) will be used. The scale consists of 13 items in total and a 5-point Likert type range is used for each item (1: strongly disagree, 5: absolutely agree). Scoring of the scale will be made according to the name of the factor. Scoring will be done in two separate groups as monitoring without being affected (Items 1, 2, 4, 7, 8, 9, 11) and Curiosity (Items 3, 5, 6, 10, 12, 13).

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Özdemir, PhD, Principal Investigator — Uludag University; Gamze Bulut, Master, Study Chair — Uludag University
Locations (1):
- Bursa Uludag University Faculty of Health Sciences, Bursa, Turkey (Türkiye)